CLINICAL TRIAL: NCT02361255
Title: Degenerative Nigrostriatal Dysfunction in Drug-induced Parkinsonism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 01481
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Secondary Parkinsonism; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease, Secondary; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Drug-induced parkinsonism: subjects with drug-induced parkinsonism
  Interventions: Other: no intervention
- antipsychotic treated non-parkinsonian control: subjects treated with antipsychotic but without parkinsonism
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Parkinson's disease (PD) and Drug-induced Parkinsonism (DIP) can be clinically indistinguishable and DIP sometimes represents "unmasking of underlying PD. The objective of this study is to determine the relationship of underlying Parkinson's disease (PD) to the incidence and clinical outcome in DIP using non-motor assessments as a marker for nigrostriatal degeneration.

Research Design: This is a nested case-control design to investigate risk factors associated with the development of DIP and persistent Parkinsonism after antipsychotic (AP) withdrawal (a potential clinical marker of underlying PD). Target enrollment is 45 subjects.

Methodology: We will examine objective olfactory function (via objective olfactory testing), other non-motor symptoms of PD (via standardized validated questionnaires), and motor findings (via clinical exam and quantitative gait analysis) in: 1) DIP patients (30 subjects) compared to AP-treated patients without Parkinsonism (15 subjects) and 2) patients with persistent Parkinsonism compared to those whose symptoms resolve in the DIP cohort followed prospectively after a change in AP treatment. Additionally, in patients where it was performed clinically, we will evaluate dopamine transporter SPECT imaging (DaTI) as a marker of nigrostriatal integrity examining the ability of qualitative and semi-quantitative analysis to distinguish between pharmacologic and degenerative Parkinsonism. We will also measure serum uric acid and Apolipoprotein A1, two putative biomarkers in early PD, and examine their relationship with clinical and radiologic status.

ELIGIBILITY:
Inclusion Criteria:

antipsychotic treated patients with or without parkinsonism

Exclusion Criteria:

parkinson's disease, dementia

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: antipsychotic treated patients with or without parkinsonism
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
normal or abnormal DAT SPECT | baseline

CONTACTS AND LOCATIONS:
Overall Officials: James Morley, Principal Investigator — PVAMC
Locations (1):
- PVAMC, Philadelphia, Pennsylvania, United States